CLINICAL TRIAL: NCT00319202
Title: A Randomized, Double Blind, Cross-Over, Placebo-Controlled Clinical Trial to Assess the Effects of Candesartan on the Carbohydrate Metabolism, of Non Diabetic, Non Hypertensive Subjects With Dysglycemia and Abdominal Obesity."ARAMIA"
Brief Title: Clinical Trial to Assess the Effects of Candesartan on the Carbohydrate Metabolism of Obese Subjects
Acronym: ARAMIA
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulties in completing the required sample size
Sponsor: Fundación Cardiovascular de Colombia (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: fcv193
Record Dates: First submitted 2006-04-26; First posted 2006-04-27 (Estimated); Last update posted 2012-11-06 (Estimated); Status verified 2012-11

CONDITIONS: Glucose Intolerance; Obesity
Keywords: Impaired fasting glucose; Abdominal obesity; HOMA; Angiotensin-receptor blocker
MeSH Terms: conditions — Glucose Intolerance; Obesity; Obesity, Abdominal | interventions — candesartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Candesartan
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Candesartan — 32 mg/d for 6 months
  Arms: 1
Drug: Placebo — Placebo administration for 6 months
  Arms: 2

SUMMARY:
Hypothesis:

The use of candesartan 16-32 mg/d for 6 months improves the carbohydrate metabolism, and decreases the plasmatic levels of adipocytokines and oxidative stress markers, in non diabetic, non hypertensive subjects with dysglycemia and abdominal obesity, and these effects are independent of the changes in arterial blood pressure.

General Objectives:

The objective is to study the impact of the treatment with candesartan in the carbohydrate metabolism and the plasmatic levels of adipocytokines and oxidative stress markers, in non diabetic, non hypertensive subjects with dysglycemia and abdominal obesity.

Study Design:

This is a randomized, double blind, cross-over, placebo-controlled, clinical trial to assess the effects of candesartan (up to 32 mg/d for 6 months), over the carbohydrate metabolism, plasma levels of adipocytokines and concentrations of oxidative stress markers in non diabetic, non hypertensive, dysglycemic and obese subjects from Colombia. The total duration of the study is 36 months.

Population:

One hundred non diabetic, dysglycemic and obese, subjects of both genders, over 18 years old, will be included. To be included subjects should have blood pressure values under 140/90 mmHg and should be receiving no antihypertensive medical treatment.

Procedures:

Subjects whom fulfill all selection criteria will be included in a run-in period of 15 days with placebo and hygiene-dietary measures (MHD) including educational, nutritional and exercise support. The patients that during this "Run in" phase have a compliance equal to or greater than 80% will be randomized to one of the two treatment groups ("Group A" receiving candesartan 16/32 mg/d for 6 months and then placebo for 6 months, or "Group B" receiving placebo during the first 6 months and then candesartan 16/32 mg/d during the last 6 months) in a 1:1 proportion by blocks of 4 subjects. Randomization will be performed by the AstraZeneca clinical department. Both groups will concurrently receive the standard treatment with MHD. Control visits will be programmed every month. Metabolic parameters, including C-reactive protein (CRP), interleukin-6 (IL-6), adiponectin, leptin, insulin, malonaldehyde and 8-isoprostanes, will be evaluated every 6 months (at the beginning and end of each treatment).

Statistical Analysis:

The analysis strategy will be performed by intention-to-treat. In a descriptive analysis, the averages and proportions will be obtained with their corresponding 95% confidence intervals for the clinically relevant variables during the baseline evaluation. In order to evaluate the differences between the groups, the Student's t test, Mann-Whitney and Fischer's exact tests will be used according to the nature of the study variables. Multiple lineal regression will be used with the purpose of comparing the treatment groups from baseline and its changes up to the 6th month of treatment.

Ethical Aspects:

The study will be conducted according to the Helsinki declaration, the good clinical practices guidelines and the Colombian legislation. Prior to entering the study, patients must sign a written informed consent that has been approved by the Institutional Ethics Committee of Fundación Cardiovascular de Colombia.

DETAILED DESCRIPTION:
Background:

During the last years, the worldwide prevalence of diabetes mellitus type II (DM2) has increased dramatically, impacting the cardiovascular morbidity and mortality. It has been estimated that more than 171 million people suffer this disease (2.8% of the worldwide population) and it's predicted that it will increase to 366 million (6.5 %) in 2030, from which 298 million will be from developing countries. Currently, in Latin America, the DM2 prevalence ranges are between 1.2% and 8%, and it is expected to increase 38% during the next 10 years, with higher levels in the urban zones.

Recently, we have demonstrated that the Colombian population with a lower abdominal circumference than those reported in Caucasian populations presented an increased risk of developed metabolic syndrome and coronary artery disease. Moreover, abdominal obesity in our population is associated with higher levels of inflammatory markers, as C-reactive protein (CRP) and proinflammatory cytokines. Nowadays, the relationship between abdominal obesity, inflammation, insulin resistance, diabetes mellitus type 2, metabolic syndrome and cardiovascular disease is a crucial aim of research, especially in populations as the Colombian, that is in high risk of being affected by the epidemic of diabetes mellitus and cardiovascular disease. The occurrence of DM2 is associated with a 2 to 4 fold increase in the risk of developing coronary disease. The diabetic patients that present unstable angina have a greater risk of developing acute myocardial infarct (AMI) and the diabetic patients with AMI have more risk of death than the non-diabetic patients. Additionally, the subjects with DM2 have an increased risk of experiencing cardiovascular events (1.5 to 3 times), and greater recurrence and mortality for these causes. The incidence and severity of the peripheral arterial disease are also increased from 2 to 4 times in diabetic patients.

The current criteria for DM2 diagnosis established by the American Association of Diabetes is a glucose level in fasting >126 mg/dl, which has been established based on the risk of suffering ophthalmic and renal micro-vascular complications with values superior to this limit. Nevertheless, several works have shown that patients with altered fasting glucose levels (≥100 mg/dl - <126 mg/dl) have an increased risk of cardiovascular morbidity and mortality.

We recently reported in Colombia, the existence of a strong association between the presence of cardiovascular risk factors and altered fasting plasma glucose, this association being greater with the presence of abnormal glucose blood levels after the glucose overload test. This association has been explained since the hyperglycemia per-se may be implicated in the development of atherosclerosis due to metabolic and structural changes at the endothelial level. At long term it may result in irreversible alterations; a "non-returning" point leading to cardiovascular complications typical of diabetes. According to these observations, our group has recently shown that patients with altered glycemia in fasting, regardless of other classic factors of cardiovascular risk, present a greater risk of coronary disease, supporting the hypothesis that the hyperglycemia leads to structural changes in the endothelial wall.

It is well known that people with insulin resistance present less vasodilatation mediated by insulin and an altered endothelium dependent vasodilatation. Additionally, it has been described that insulin causes a physiologic vasodilatation in the skeletal muscle of healthy subjects, an effect that is blocked in insulin-resistance obesity. In our population, we find that obesity, hypercholesterolemia and diabetes are related with a flow-mediated vasodilatation reduction. The endothelial dysfunction is strongly related with the insulin resistance syndrome. At the same time, the endothelial dysfunction worsens the resistance to insulin, increases the vascular reactivity and predisposes to cardiovascular disease. It has been proposed that the vasodilator effect of the insulin is primarily due to a greater expression of mRNA for endothelial nitric oxide synthase (eNOS) due to a probable increase of the transcriptional rate. There are elements to support the fact that this activity is modulated by C-kinase protein (PKC). The inhibition of PKC increases the mRNA levels for eNOS. Prolonged incubation of endothelial cells with a selective inhibitor of the PKC beta isoform increase the mRNA levels of eNOS. This observation may have important clinical implications since the PKC activation in the vasculature of diabetic subjects in alteration of the vascular wall. The existing relationship between endothelial dysfunction and insulin resistance is dependent on multiple factors. Obesity generates an alteration of the endothelial function in the metabolically active capillary bed, altering the lipase lipoprotein (LPL) that is linked to the endothelium by glycosaminoglycans. The ultimate loss of these caused by aggressive factors such as smoking and oxygen free radicals, alters the endothelial function and also impairs the action of the LPL causing hypertriglyceridemia which is an insulin resistance factor. At the same time, the alteration of endothelial function in the capillary beds reduces the interstitial flow, carrying less insulin or delaying its delivery to the muscular tissue. Additionally, it has been proposed that there is less surface of endothelium functionally normal in the vessels that are irrigating the skeletal muscle. It has also been shown that hyperinsulinemia predicts the appearance of atherosclerosis and cardiovascular events, independently of other risk factors.

The increase of adipocytes at the abdominal level is directly related with a condition of insulin resistance and hyperinsulinism. The hyperinsulinemia promotes the release of free fatty acids by the adipocyte and its later hepatic transformation to oxidized LDL, which have a great atherogenic potential. Also, the abdominal adipocytes in response to the increase of free fatty acids, oxidized LDL or any other non-well defined metabolic factor increase the production and release of proinflammatory cytokines such as the tumor necrosis factor alpha (TNF-α) and interleukin-6 (IL-6), which have shown to be able to reduce the expression and activity of the nitric oxide synthase (eNOS) in human cultivated umbilical endothelium cells, suggesting that this could be the mechanism by which the abdominal obesity is related with endothelial dysfunction. In this sense, we have recently demonstrated that in cultured endothelial cells, the angiotensin II, through receptor AT1, stimulates the TNF-α production, which at the same time activates the metalloproteinase 2, enzyme which induces changes in the endothelium structure and in the stability of the atherosclerotic plaque. This effect of angiotensin II is mediated by the AT1 receptor, since we have shown that the CANDESARTAN inhibited the production of TNF-α induced by Angiotensin II.

The increase in the production and storage of free fatty acids may be the mechanism by which angiotensin II relates with the development of insulin resistance. It has been demonstrated that the elevated levels of free fatty acids induce insulin resistance through the inhibition of the transport and phosphorylation of glucose at a muscular level, followed by a reduction of the glycogen synthesis and glucose oxidation. Additionally, it has been suggested that free fatty acids may interfere in the stimulation of insulin in the GLUT 4 and hexokinase activity. Also, angiotensin II has a stimulating effect on the transcription rate of the ob gene in human adipocytes. The ob gene is in charge of codifying the leptin protein, which inhibits the appetite and regulates the thermogenesis. The chronic and sustained increase in leptin levels leads to a leptin-resistance condition, a condition in which the hormone loses its physiological actions. The increase in the leptin levels produces a greater expression of UPC 2 (Uncoupling protein 2) in an action mediated by Peroxisome Proliferator-Activated Receptors (PPARs), which interferes with the mitochondrial respiration chain in the pancreatic beta cells, getting to a reduction in the ATP generation and blocking the first peak of insulin secretion. This offsetting mechanism seems to be opposed to the insulin's lipogenic effect and avoids greater lipid storage. Unfortunately, the derived consequences of this alteration in the insulin secretion are a lower efficacy to maintain the euglycemia and to maintain a glucidic homeostasis. On the other hand, the hyperleptinemia, by mediating the sympathetic activity and increasing the sodium renal resorption, leads to the increases of blood pressure, which adds to the greater expression of the angiotensinogen produced by hypertrophied lipid cells. These cells generate angiotensin II to activate the adipocyte differentiation and to regulate the fat storage in response to nutritional changes.

Recently, some clinical trials have demonstrated that the angiotensin converting enzyme inhibitors (ACEIs) and ARA II, reduce the risk of presenting new cases of DM2 as compared with other antihypertensive therapies. However, no clinical trials have addressed specifically the study of the effects of the ARA II in the improvement of the dysglycemia and in the prevention of the diabetes type 2. Additionally, the treatment with ACEI and ARA II has shown to improve the resistance to peripheral insulin both in animal models and clinical studies. The mechanism by which the renin-angiotensin-aldosterone system blockade has a beneficial effect on the responsiveness to insulin has not been totally cleared. In obese Zucker-type rats, it was demonstrated that the chronic treatment with a selective ARA II receptor produced a significant increase in the GLUT 4 transporter expression in skeletal muscle and a reduction in the concentrations of plasma fatty acids associated with an improvement of the responsiveness to insulin.

Although the mechanisms are still speculative, the beneficial effects of the renin-angiotensin system blockade, demonstrated in several studies such as HOPE, LIFE, VALUE, on the responsiveness to insulin and in the prevention of the development of new cases of DM2, suggest that angiotensin II produced in the adipocytes of obese subjects is associated to the insulin resistance syndrome and supports the execution of clinical trials oriented to establish the beneficial effect of ARA II in the prevention of DM2 in susceptible individuals coming from populations at high risk of developing CVD and diabetes mellitus, as the Colombian one.

Hypothesis:

In non-diabetic non-hypertensive subjects with dysglycemia and abdominal obesity:

The treatment with candesartan 16/32 mg/d during 6 months improves carbohydrate metabolism measured by HOMA insulin sensibility index, oral glucose tolerance Test (OGTT), fasting plasma glucose levels, and glycosylated hemoglobin (HbA1c).

The effects of the treatment with candesartan over carbohydrate metabolism is related to a reduction in the plasma concentration of adipocytokines such as IL-6, CRP, Leptin and Adiponectin; and oxidative stress markers such as plasma concentrations of Malonaldehyde and urinary concentration of 8-Isoprostanes.

These effects over carbohydrate metabolism, inflammatory adipocytokines or oxidative stress markers are independent of changes over arterial blood pressure.

Study Objectives:

General Objectives:

To study the impact of the treatment with candesartan over the carbohydrate metabolism, inflammatory adipocytokines and levels and oxidative stress markers in non-diabetic non-hypertensive subjects with dysglycemia and abdominal obesity.

Specific Objectives:

In non-diabetic non-hypertensive subjects with abdominal obesity and dysglycemia:

To establish the impact of the treatment with candesartan (16/32 mg/d) in the carbohydrate metabolism assessed through the HOMA index, fasting glucose plasma levels, OGTT, and HbA1c levels.

To study the effects of candesartan 16/32 mg/d during 6 months over fasting plasma levels of adipocytokines such as Leptin, Adiponectin, IL-6 and CRP.

To determine if the treatment with candesartan (16/32 mg/d during 6 months) decreases the concentration of oxidative stress markers such as plasma levels of malonaldehyde and urinary levels of 8-Isoprostanes.

To determine if the effects of candesartan on the carbohydrate metabolism, adipocytokines and oxidative stress marker concentrations, are independent of its effect upon the blood pressure.

Study Design:

A randomized, double blind, placebo-controlled, cross-over clinical trial, to assess the effects of candesartan (16/32 mg/d during 6 months) over metabolic, oxidative, and inflammatory parameters, in non-diabetic non-hypertensive subjects with dysglycemia and abdominal obesity.

Study treatments:

Treatment A: Candesartan 16 mg (one tablet per day) taken with breakfast during 4 weeks, depending on the subject's tolerance the dosage will be increased to 32 mg/d (two tablets) during the next 20 weeks.

Treatment B: Placebo tablets administered similarly to treatment A (one tablet during 4 weeks and then 2 tablets per day during the next 20 weeks).

All subjects will be included in a hygiene-dietary measures program (MHD; educational, nutritional and exercise support) during the study.

Study groups:

The study embraces two arms

Group 1: Will receive treatment A first during the first 24 weeks and then treatment B during the last 24 weeks.

Group 2: Will receive treatment B during the first 24 weeks and then treatment A during the last 24 weeks.

Population:

The study is going to be integrated by non-diabetic non-hypertensive subjects of both genders, older than 18 years with abdominal obesity and dysglycemia .

Abdominal obesity is defined as a waist diameter greater than 90 cms in men and 80 cms in women.

Dysglycemia is defined as having plasma glucose levels in fasting between 100 and 125 mg/dL and/or on glucose tolerance test at 2 hours between 140 mg/dL and 200 mg mg/dL.

Size of sample:

The size of the sample was estimated considering a crossover, clinical trial design and following the proposal by Hills and Armitage accepting a type I error of 0.05, a power of 90%, and assuming a difference of 20% in the HOMA index after 6 months of treatment with candesartan (3 to 2.4) and a maximum standard deviation of 1.5, sample size of 84 subjects was estimated. By adjusting the rate of losses of 8%, the final sample size is 100 subjects (50 in each group).

This sample size ensures a power of 90% to detect differences in the fasting glycemia of at least 8mg/dL (0.44mmol/L), with a standard deviation (SD) of 20mg/dL. (1.1mmol/L) or a difference of 14mg/dL (0.77mmol/L) in the 2 hours post load glycemia SD of 40mg/dl (2.2mmol/L).

Statistical Analysis:

The study is fundamentally set forth as an efficacy study on the prevention of the development of diabetes mellitus and on the changes of the carbohydrate metabolism. The averages and proportions with their corresponding 95% confidence intervals for clinically relevant variables measured during the baseline evaluation will be obtained in a descriptive analysis. In order to evaluate the presence of differences between the groups, the Student's t test, the Mann-Whitney test, the CHI2 test or the Fisher´s exact test according to the variable under study will be used. A Linear multiple regression will be used with the purpose of comparing the treatment groups from baseline and its changes up to month end 6 of each treatment. The possibility of performing adjustments by required baseline parameters and risk factors and prior treatment in each one of the treatment groups is considered.

The analysis will be performed by the intention-to-treat approach. A p value under 0.05 will be considered as statistically significant.The primary endpoint for analysis will be made on the change in HOMA index value, baseline glucose, and post-charge glucose plasma levels. The secondary endpoint for analyses will include the possible changes in serum insulin, leptin and adiponectin, inflammatory markers and oxidative stress markers .

Treatment safety register and analysis will be made through the clinical review and statistics of the adverse events reported.

Safety Committee and Events Assignation Committee:

A safety and events assignation committee will be created, according to the Harmonized Tripartite Guidelines of the International Conference of Harmonization for Good Clinical Practices.

Ethical Aspects:

The clinical trial will be conducted according to the Helsinki's Declaration, Good Clinical Practice Guidelines and the Colombian legislation (Resolution 8430-93 of the Ministry of Health). The patient will provide written informed consent in a form designed for such a purpose.

The information generated by the study will be confidential and strictly used for the purposes stipulated within the protocol.

Finally, the patient may refuse to continue participating in the study at any moment after providing his/her consent. The study will be approved by the FVC ethics committee. All assessments will be performed by trained staff. The blood samples will be collected in aseptic conditions by an expert bacteriologist.

Study Timeline:

The study period will be 36 months. The initiation will be defined by the project's financial approval.

ELIGIBILITY:
Inclusion Criteria:

The subjects that fulfill the following inclusion criteria will be eligible to participate in the study:

* Men and women older than 18 years of age.
* Waist perimeter > 90 cm in males or > 80 cm in females
* Have plasma glucose levels in fasting between 100 and 125 mg/dL and/or on glucose tolerance test at 2 hours > 140 mg/dL and < 200 mg/dL.
* Having a treatment compliance of over 80% at the end of the run-in phase.
* All women with childbearing potential must have a secure contraceptive method. A secure method will be considered as sterilization by surgical methods, postmenopausal condition with an age greater than 45 years and a menopausal period equal to or greater than two years. In premenopausal women, the use of two barrier contraceptive methods including 1 month after the conclusion of the active phase of study treatment.

Exclusion Criteria:

Individuals with any of the following characteristics will be excluded:

* Prior diagnosis of type 1 or 2 diabetes mellitus, chronic or acute renal insufficiency, coronary disease clinically evident (acute myocardial infarction, chest angina, myocardial revascularization) or cardiac insufficiency, or history of prior cardiovascular events (AMI, CVD, or CABG).
* Significant chronic disease (terminal stage cirrhosis or hepatic disease or cancer) that affects the survival of patients at 12 months.
* Chronic inflammatory diseases of obesity (lupus erythematosus, rheumatoid arthritis, etc.)
* Infectious acute or chronic processes of any etiology with an occurrence within the 4 weeks prior to the beginning of the study.
* Use of steroid hormones or NSAIDs 1 month prior to the beginning of the study.
* The patient is participating in a program or under treatment to lose weight during the 8 weeks prior to the study entry.
* The patient requires (for any circumstance) treatment with immunosuppressive agents.
* Has participated in a clinical trial in the 8 weeks prior to the study entry.
* At the study entry, the patient is considering the possibility of a surgical procedure during the next 12 months.
* History of severe chronic gastritis or any condition of the gastrointestinal tract that may affect the absorption and/or distribution of any drug administered orally.
* Alteration of the hepatic function tests. The maximum value for ALT or AST will be considered as > 2 times the upper normal limit.
* Triglycerides > 600 mg/dl.
* History of the use of psychoactive drugs or abuse of alcohol.
* Positive pregnancy test in the screening visit.
* Concomitant treatment with any other antihypertensive drug.
* Contraindication to receive treatment with candesartan.
* Pathological alterations of aortic or mitral cardiac valves (stenosis or insufficiency) or hypertrophic cardiomyopathy.
* Denial to sign informed consent, or any mental condition that makes the patient part of a susceptible population

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2006-06; Primary Completion 2010-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Changes in HOMA index value | 6 months after beginning the treatment

SECONDARY OUTCOMES:
Changes in serum insulin, leptin and adiponectin, inflammatory markers and oxidative stress markers | 6 months after beginning the treatment
Changes in baseline glucose, and post-charge glucose plasma levels | 6 months after beginning the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G Garcia Gomez, MD, PhD, Principal Investigator — Research Institute/Fundación Cardiovascular de Colombia; Vicente Lahera, PhD, Study Chair — Departamento de Fisiologia/Universidad Complutense de Madrid; Federico A Silva, MD, Study Chair — Research Institute/Fundación Cardiovascular de Colombia; Gustavo Marques, MD, Study Chair — Research Institute/Fundación Cardiovascular de Colombia
Locations (1):
- Fundación Cardiovascular de Colombia, Floridablanca, Santander Department, Colombia

REFERENCES:
- [Derived] Lopez-Jaramillo P, Pradilla LP, Lahera V, Sieger FA, Rueda-Clausen CF, Marquez GA. A randomized, double blind, cross-over, placebo-controlled clinical trial to assess the effects of Candesartan on the insulin sensitivity on non diabetic, non hypertense subjects with dysglyce mia and abdominal obesity. "ARAMIA". Trials. 2006 Sep 7;7:28. doi: 10.1186/1745-6215-7-28. PMID 16959033
- See also: Official web site of the Fundacion Cardiovascular de Colombia — http://www.fcv.org